CLINICAL TRIAL: NCT06589596
Title: A Phase 1a/b Study Investigating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of PRMT5 Inhibitor BGB-58067 Alone and in Combination With Anticancer Agents in Patients With Advanced Solid Tumors
Brief Title: An Investigational Study of BGB-58067 As a Single Agent and in Combination With Anticancer Agents in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-58067-101; 2024-515307-19-00 (EU CTIS Number); CTR20244451 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor
Keywords: advanced solid tumor; BGB-58067; MTAP deficiency; BG-89894

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1a: BGB-58067 Monotherapy Dose Escalation and Safety Expansion (Experimental): Sequential cohorts of increasing dose levels of BGB-58067 as monotherapy will be evaluated.
  Interventions: Drug: BGB-58067
- Phase 1a: BGB-58067 + BG-89894 Combination Therapy Dose Escalation (Experimental): Sequential cohorts of increasing dose levels of BGB-58067 in combination with BGB-89894 will be evaluated.
  Interventions: Drug: BGB-58067; Drug: BG-89894
- Phase 1a: BGB-58067 + Standard of Care Combination Therapy Dose Escalation (Experimental): Sequential cohorts of increasing dose levels of BGB-58067 in combination with standard of care therapy will be evaluated.
  Interventions: Drug: BGB-58067; Drug: Standard of Care Therapy
- Phase 1b: Dose Expansion and Optimization (Experimental): Recommended Dose(s) for Expansion (RDFE[s]) of BGB-58067 alone, in combination with BG-89894, and in combination with standard of care therapy will be evaluated for selected indications and regimen(s) based on emerging data.
  Interventions: Drug: BGB-58067; Drug: BG-89894; Drug: Standard of Care Therapy

INTERVENTIONS:
Drug: BGB-58067 — Planned doses administered on specified days per protocol.
Drug: BG-89894 — Planned doses administered on specified days per protocol.
  Arms: Phase 1a: BGB-58067 + BG-89894 Combination Therapy Dose Escalation; Phase 1b: Dose Expansion and Optimization
Drug: Standard of Care Therapy — Administered in accordance with relevant local guidelines and/or prescribing information.
  Arms: Phase 1a: BGB-58067 + Standard of Care Combination Therapy Dose Escalation; Phase 1b: Dose Expansion and Optimization

SUMMARY:
This is an open-label, multicenter, first-in-human dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary antitumor activity of BGB-58067 alone, in combination with BG-89894, and in combination with standard of care therapy in participants with advanced solid tumors and with methylthioadenosine phosphorylase (MTAP) deficiency.

DETAILED DESCRIPTION:
BGB-58067 is a new drug designed to target a specific protein called protein arginine methyltransferase 5 (PRMT5). This protein is involved in many cell activities and can promote cancer growth when it is overactive. High levels of PRMT5 are linked to poor outcomes in several types of cancer.

This new study will check how safe and helpful a potential anticancer drug called BGB-58067 is. This drug will be tested alone, in combination with BG-89894, and in combination with standard of care therapy in participants with advanced solid tumors and with MTAP deficiency.

Note: Our company, previously known as BeiGene, is now officially BeOne Medicines. Because some of our older studies were sponsored under the name BeiGene, you may see both names used for this study on this website.

ELIGIBILITY:
Inclusion Criteria:

* Participants must sign the ICF and be capable of giving written informed consent
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 or Karnofsky Performance Scale (KPS) ≥ 70
* Life expectancy ≥ 3 months
* Evidence of homozygous loss of MTAP or lost MTAP expression in the tumor tissue
* Able to provide tumor sample to meet the minimum tissue requirement for central MTAP deficiency testing
* Participants with histologically or cytologically confirmed advanced, metastatic, or unresectable solid tumors, whose diseases have progressed or recurred after receiving standard systemic therapy or radiotherapy, or for whom standard systemic therapy is not available or tolerated, or would be unlikely to tolerate or derive clinically meaningful benefit from appropriate standard treatment in the opinion of the investigator; participants with advanced, metastatic, or unresectable solid tumors who have not received prior systemic treatment or have received one cycle of standard-of-care therapies will be enrolled in selected cohorts
* Adequate organ function

Exclusion Criteria:

* Prior treatment with any methylthioadenosine (MTA)-cooperative PRMT5 inhibitor or methionine adenosyltransferase 2a (MAT2A) inhibitor
* Active leptomeningeal disease or symptomatic spinal cord compression
* Uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage
* Any malignancy ≤ 2 years before first dose of study drug except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively
* Significantly impaired pulmonary function
* Clinically significant infections
* Serologically active hepatitis B or C infection
* Known HIV infection. Participants with treated HIV infection may be included in Phase 1b if they meet certain criteria
* High cardiovascular risk factors
* QTcF > 470 ms based on the screening triplicate 12-lead ECG records and/or a history of additional risk factors for torsade de pointes (eg, heart failure, hypokalemia, or a family history of Long QT Syndrome)
* Toxicities (because of prior anticancer therapy) that have not recovered to baseline or stabilized
* Participants who are unable to swallow or with disease/procedure significantly affecting gastrointestinal function
* Female participants who are pregnant or are breastfeeding
* Concurrent participation in another therapeutic clinical study (participation in observational or noninterventional studies is allowed)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants with Adverse Events and Serious Adverse Events | From first dose of the study drug(s) to 30 days after the last dose or initiation of a new anticancer therapy, whichever occurs first (approximately 13 months)
  Number of participants with AEs and SAEs, including findings from physical examinations, electrocardiograms (ECGs), and laboratory assessments.
Phase 1a: Number of Participants with Adverse Events that meet Dose-Limiting Toxicity (DLT) criteria | Approximately 1 month
Phase 1a: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of BGB-58067 alone, in combination with BG-89894, and in combination with standard of care therapy | Approximately 1 month
  MTD is defined as the highest dose evaluated for which estimated toxicity rate is the closest to the target toxicity rate. MAD is defined as the highest dose administered if MTD is not reached.
Phase 1a: Recommended Dose(s) for Expansion (RDFE[s]) of BGB-58067 alone, in combination with BG-89894, and in combination with standard of care therapy | Approximately 13 months
  RDFE of BGB-58067 alone, in combination with BG-89894, and in combination with standard of care therapy will be determined based upon the MTD or MAD.
Phase 1b: Recommended Phase 2 Dose (RP2D) of BGB-58067 alone, in combination with BG-89894, and in combination with standard of care therapy | Approximately 2 years
  RP2D established from Phase 1a for BGB-58067 alone, in combination with BG-89894, and in combination with standard of care therapy for administration in selected tumor types.
Phase 1b: Objective Response Rate (ORR) | Approximately 2 years
  ORR is defined as the percentage of participants with confirmed complete response (CR) or partial response (PR), as assessed by the investigator.

SECONDARY OUTCOMES:
Phase 1a: Objective Response Rate (ORR) | Approximately 2 years
  ORR is defined as the percentage of participants with confirmed CR or PR, as assessed by the investigator.
Phase 1a and 1b: Maximum observed plasma concentration (Cmax) of BGB-58067 | Approximately 2 months
Phase 1a and 1b: Minimum observed plasma concentration (Cmin) of BGB-58067 | Approximately 9 months
Phase 1a and 1b: Time to reach maximum observed plasma concentration (Tmax) of BGB-58067 | Approximately 2 months
Phase 1a and 1b: Apparent oral clearance (CL/F) for BGB-58067 | Approximately 2 months
Phase 1a and 1b: Half-life (t1/2) of BGB-58067 | Approximately 2 months
Phase 1a and 1b: Area under the concentration-time curve (AUC) of BGB-58067 | Approximately 2 months
Phase 1a and 1b: Apparent volume of distribution (Vz/F) for BGB-58067 | Approximately 2 months
Phase 1a and 1b: Accumulation ratio (AR) for BGB-58067 | Approximately 2 months
Phase 1a and 1b: Plasma concentrations of BGB-58067 | Approximately 9 months
Phase 1a and 1b: Duration of Response (DOR) | Approximately 2 years
  DOR is defined as the time from the first determination of an objective response until first documentation of progression or death, whichever occurs first, as assessed by the investigator.
Phase 1a and 1b: Disease Control Rate (DCR) | Approximately 2 years
  DCR is defined as the percentage of participants with best overall response of a CR, PR, and stable disease, as assessed by the investigator.
Phase 1b: Number of Participants with AEs and SAEs | From first dose of the study drug(s) to 30 days after the last dose or initiation of a new anticancer therapy, whichever occurs first (approximately 13 months)
  Number of participants with AEs and SAEs, including findings from physical examinations, electrocardiograms (ECGs), and laboratory assessments.
Phase 1b: Progression-Free Survival (PFS) | Approximately 2 years
  PFS is defined as the time from the date of the first dose of study drug to the date of first documentation of progressive disease assessed by investigator or death, whichever occurs first, as assessed by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (47):
- United States (9):
  - Usc Norris Comprehensive Cancer Center (Nccc), Los Angeles, California
  - Adventhealth, Celebration, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Nyu Langone Health, New York, New York
  - Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
  - Next Dallas, Irving, Texas
  - Next Virginia, Fairfax, Virginia
- Australia (4):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- China (21):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital Wuxiang Branch, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai East Hospital Branch Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Centerpudong, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang, Taizhou, Zhejiang
- Rigshospitalet, Copenhagen, Denmark
- France (4):
  - Centre de Lutte Contre Le Cancer Institut Bergonie, Bordeaux
  - Institut Curie Paris, Paris
  - Institut de Cancerologie de Louest, Saint-Herblain
  - Institut Gustave Roussy, Villejuif
- South Korea (4):
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, SongpaGu, Seoul Teugbyeolsi
- Spain (4):
  - Hospital Universitario Vall Dhebron, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Start Madrid Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Hm Madrid Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/